CLINICAL TRIAL: NCT06005844
Title: Validation of the Performance of the French Version of the Cerebellar Cognitive-Affective Syndrome Scale (CCASS) as a Screening Test for Cerebellar Cognitive-affective Syndrome: a National Multicenter Study
Acronym: CCASS-FR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GHRMSA 1228
Record Dates: First submitted 2023-08-07; First posted 2023-08-23 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Cerebellar Cognitive-affective Syndrome
Keywords: Schmahmann syndrome; Cerebellar cognitive-affective syndrome; Screening
MeSH Terms: conditions — Cerebellar Cognitive Affective Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adults with a cerebellar damage (Other)
  Interventions: Diagnostic Test: Cerebellar Cognitive-Affective Syndrome Scale

INTERVENTIONS:
Diagnostic Test: Cerebellar Cognitive-Affective Syndrome Scale — The CCASS will be administered by a neuropsychologist starting with version 1A. An alternative version (1B, 1C or 1D) will also be administered. An interval of approximately 30 minutes should be observed between the two administrations. In order to assess the inter-rater reliability of the scale, a second neuropsychologist will be present in the room and will independently evaluate (i.e., blind to his/her colleague's rating) patient's responses. The choice of alternative version (i.e., 1B, 1C, or 1D) will be randomized.

SUMMARY:
The primary objective of the study is to assess the performance of the French version of the Cerebellar Cognitive-Affective Syndrome Scale (CCASS) as a screening test for cerebellar cognitive-affective syndrome.

The primary endpoint will be the sensitivity of version 1A of the French scale. The result will be considered positive if the patient fails at least one of the scale's subtests. The diagnosis of a cerebellar cognitive-affective syndrome will be made on the basis of a pathological score in the executive, language, visuospatial or psychoaffective domains of the neuropsychological evaluation (gold standard).

DETAILED DESCRIPTION:
Secondary objectives:

1. To determine the other accuracy measures for version 1A of the French CCAS scale;
2. To determine the performance indices (i.e., sensitivity, specificity) of French versions 1B, 1C and 1D of CCAS scale;
3. To determine the performance indices of versions 1A, 1B, 1C, and 1D of CCAS scale when positivity is defined by ≥ 2 or ≥ 3 failed subtests, respectively;
4. To evaluate the consistency of results from versions 1B, 1C and 1D compared with version 1A;
5. To assess the inter-rater reliability of the different versions of the French scale;
6. To assess the learning effect on version 1A of the French scale in the subgroup of patients included at Mulhouse hospital;
7. To measure the time taken by patients to complete version 1A of the French scale.

   Conduct of research:

   The study will take place in the following french centers: GHRMSA - Hôpital Emile Muller (Mulhouse), AP-HP - Hôpital Pitié-Salpêtrière (Paris), CHRU Nancy - Hôpital Central (Nancy), Hôpitaux civils de Colmar (Colmar).

   - V0 Screening: The protocol will be proposed to all eligible patients by the investigator.

   - V1 Inclusion visit and CCASS test: The inclusion visit will be scheduled on the date of the patient's next follow-up medical appointment.

   The CCASS will be administered by a neuropsychologist starting with version 1A. An alternative version (1B, 1C or 1D) will also be administered. An interval of approximately 30 minutes should be observed between the two administrations. In order to assess the inter-rater reliability of the scale, a second neuropsychologist will be present in the room and will independently evaluate (i.e., blind to his/her colleague's rating) patient's responses, without directly interfering in the administration of the scale.

   The choice of alternative version (i.e., 1B, 1C, or 1D) will be randomized.

   - V2 Gold standard: Within 7 days of completing CCASS, a complete neuropsychological assessment will be carried out by a third neuropsychologist, blinded to the results of the scale.

   - V3 Re-testing of version 1A of CCASS: In the subgroup of patients included at Mulhouse hospital, a second administration of version 1A of CCASS will be carried out by one of the two neuropsychologists who carried out the V1 visit.

   V3 will be scheduled 80 to 100 days after V1..

ELIGIBILITY:
Inclusion criteria :

* French speaking
* Acquired lesion or predominantly degenerative cerebellar pathology of any etiology
* Affiliated or beneficiary of a social security scheme
* Written informed consent

Non-inclusion criteria:

* History or progressive pathology of the central nervous system other than cerebellar disease
* Chronic ethylic patient with active consumption, or alcohol withdrawal of less than three months
* Use of other toxic substances
* Blind or severely visually impaired patient
* Deaf or severely hearing-impaired patient unable to understand instructions
* Mute patient
* Patient deprived of liberty or under legal protection

Secondary exclusion criteria :

- Patients with incomplete French scale and/or neuropsychological assessment will be replaced.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the 1A French version of the cerebellar cognitive-affective syndrome scale | Up to 7 days

SECONDARY OUTCOMES:
Specificity of the 1A French version of the cerebellar cognitive-affective syndrome scale | Up to 7 days
Sensitivity and specificity of the 1B, 1C and 1D French versions of the cerebellar cognitive-affective syndrome scale | Up to 7 days
Sensitivity and specificity measured on the different versions of CCASS when a positive result is defined by ≥ 2 or ≥ 3 failed subtests respectively. | Up to 7 days
Concordance between the total raw score of version 1A and the total raw score of versions 1B, 1C, 1D, evaluated graphically using the Bland and Altman method | Day 1
Inter-rater agreement measured on the total raw score of the different versions of the French scale by calculating the intraclass correlation coefficient and using the Bland and Altman method | Day 1
Time to complete version 1A of the French scale | Day 1
Total raw score on version 1A at V3 | Up to 100 days
  The learning effect will be assessed in the subgroup of patients included at Mulhouse hospital. Comparison of the total raw score on version 1A at V1 and the total raw score on version 1A at V3 will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- GHRMSA, Mulhouse, Haut-Rhin, France

IPD SHARING:
Plan to Share IPD: No